CLINICAL TRIAL: NCT05813743
Title: How Accurate is Three Dimensional Ultrasonography in Prenatal Detection of Urinary Bladder Wall Involvement in Abnormally Invasive Placenta at 3rd Trimester of Pregnancy ?
Brief Title: Detection of Urinary Bladder Wall Involvement in Abnormally Invasive Placenta (AIP) by 3D Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Abnormally invasive placenta
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Placenta Accreta
Keywords: Abnormally invasive placenta; 3D ultrasound
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant in 3rd trimester with abnormally invasive placenta (Other)
  Interventions: Diagnostic Test: 3 dimensional ultrasound

INTERVENTIONS:
Diagnostic Test: 3 dimensional ultrasound — Detect the accuracy of 3D ultrasonography in prenatal detection of bladder wall involvement in abnormally invasive placenta (AIP) at 3rd trimester of pregnancy .

SUMMARY:
In the last three decades , the raise in cesarean delivery rates has led to a massive increase in the incidence of the abnormally invasive placenta .Complete separation of the abnormally invasive placenta is very difficult and usually fails and this may leads to life threatening hemorrhage and other morbidities e.g injury of the urinary tract.

Antenatal diagnosis of the extent of the myometrial involvement may help in the anticipation and the planning of management eg: to proceed a conservative management or cesarean hysterectomy in case of extensive myometrial involvement . Three dimensional (3D) power Doppler ultrasound now represents a turning point for diagnosis the abnormal placentation .

DETAILED DESCRIPTION:
Our study aimes to detect the accuracy of 3D ultrasonography in prenatal detection of urinary bladder wall involvement in abnormally invasive placenta (AIP) at 3rd trimester of pregnancy .

All patients will be subjected to the following:

1-Written informed consent after explaining the aim of the study, procedure and possible hazards.

2-History taking includes full obstetric history, medical and surgical history. 3-Relevant physical examination.

* In all cases, detailed transabdominal and transvaginal examinations of the placenta, uterus and pelvis will be performed within 48 hours before surgery will be done by ultrasound equipment type (GE Voluson E10).
* During the ultrasound examination the following criteria will be studied:

  1. Placental localization and determining placental extension : The placenta will be recorded as low lying when the edge is 0.5-2 cm from the internal os of the uterine cervix. When the placenta is <0.5 cm from the internal os or completely covering it, it will be defined as placenta previa (marginal or complete respectively).
  2. The criteria suggested by the European working group on Abnormally invasive placenta (EW-AIP)25 which include:

     * Loss of clear zone in the myometrium under the placental bed.
     * Myometrial thinning to less than 1 mm.
     * Intra-placental lacunae which are large and irregular.
     * Bladder wall interruption or loss.
     * Placental bulge or focal exophytic mass extending beyond the serosa of the uterus.
* Color Doppler images:

  -- Uterovesical hypervascularity between placenta and posterior wall of the bladder.
  * Bridging vessels across the myometrium and beyond uterine serosa.
  * Sub-placental hypervascularity.
  * Lacunae feeder vessels with high velocity.
* The results of 3D ultrasound will be compared with the results of histopathological examination of the retrieved specimens in cases of cesarean hysterectomy or partial myometrial resection or with the operative finding of spontaneous and complete placental separation at laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Previous cesarean deliveries
* Gestational age (GA)> or= 28 weeks
* Low lying placenta previa totally or partially covering the internal os with lateral +/- anterior wall extension diagnosed as placenta accreta spectrum (PAS) disorders by 3D ultrasound

Exclusion Criteria:

* Patient's refusal to participate
* Multifetal pregnancies
* Gestational age< 28 weeks.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of 3 dimensional ultrasound in detection of urinary bladder invasion in patients with abnormally invasive placenta | 6 months
  The sensitivity and specificity of three dimensional ultrasound in the diagnosis of bladder wall invasion in patients with abnormally invasive placenta

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided